CLINICAL TRIAL: NCT01409044
Title: The Effect of Music Listening on the Amount of Opioids Used in Surgical Intensive Care Patients
Brief Title: Effect of Music on Pain and Anxiety After Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 110201; 11-CC-0201
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08-08

CONDITIONS: Postop Adult ICU Patients
Keywords: Patient-Controlled Analgesia (PCA); Music Listening; Opioids; Post Surgical Intensive Care Patient; Patient-Controlled Analgesia
MeSH Terms: interventions — Music Therapy

ARMS (1):
- Music (Experimental): Research participant listened to music
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — Music listening for the treatment group. Music is from MusicCure selection "Dreams". Outocmes are compared to control group who receives no music. Subjects are randomized Post-operatively.

SUMMARY:
Background:

- Studies have shown that listening to music can decrease pain and anxiety. Following surgery, patients in intensive care units (ICUs) often need drugs to treat their pain and anxiety. But these drugs can cause side effects such as low blood pressure and confusion. If listening to music can help lower pain and anxiety levels, less medication might be needed and these side effects could be avoided.

Objectives:

- To determine the effects of music on patient pain and anxiety in the first few days after surgery.

Eligibility:

- Individuals at least 18 years of age who are scheduled to have surgery that requires a 24-48-hour stay in intensive care afterward.

Design:

* All participants will be screened with a medical history before having surgery.
* Participants will be divided into two groups: one group will listen to music after surgery, and the other will not.
* Before surgery, participants will answer questions about their pain and anxiety levels. They will also be shown how to control the device that lets them administer their own pain medication after surgery.
* Following surgery, all participants will be transferred to the ICU and will answer the same questions about pain and anxiety levels.
* The music group will listen to a specially created CD of instrumental music for about 50 minutes, four times a day. The standard group will not listen to this music. All other treatments will be the same in both groups. Both groups will continue to answer the same questions about pain and anxiety levels.
* Participants will have a final 15- to 20-minute interview after leaving the ICU. They will answer questions about the ICU stay and (for those in the music listening group) the music.

DETAILED DESCRIPTION:
Background:

* Listening to music is a common human activity. Music listening has been associated with decreased pain scores, increase in attentiveness and decrease in anxiety scores. Recently, with interest in holistic and complementary and alternative therapies, there has been increased awareness of the potential positive health effects of music listening.
* Inadequate pain management remains common especially in postoperative patients. Acute perioperative pain affects over 46 million Americans every year.
* As music is processed by the limbic system, enkephalins and endorphins are released. These substances are natural occurring opioids, suggesting music may decrease patient s requirements for opioids.

Primary Objective:

To determine the effects of music listening on the amount of opioids delivered postoperatively to adult ICU patients via patient-controlled analgesia (PCA) during the first 48 hours.

Secondary Objective:

To determine the effects of music listening on pain and anxiety scores experienced by adult surgical patients during the first 48 hours postoperatively in the ICU.

Eligibility:

-All adult patients (18 years of age or greater) who are scheduled for surgery that have an anticipated ICU stay of 24-48 hours.

Design:

The design is a two-group randomized controlled trial. The two groups are:

* Treatment -Music group - intervention music delivered for approximately 50 minutes 4 times a day
* Control - Standard care

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult surgical patients hospitalized in the NIH, Clinical Center (CC) who have an anticipated ICU stay of 24-48 hours postoperatively and the planned postoperative pain management schema includes opioids delivered via intravenous or epidural PCA device.
* General surgery, urology and thoracic surgery patients
* Oriented to person, time and place
* Age greater than or equal to 18 years
* Understands and speaks English or Spanish

EXCLUSION CRITERIA:

* Scheduled for a neurosurgical procedure
* Hearing or visually Impaired
* Diagnosed with General Anxiety Disorder (GAD) or patients who score greater than or equal to 15 on the GAD-7 screening instrument.
* Speaks language other than Spanish or English
* Intubated for greater than 4 hours post-operatively

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-06-17; Primary Completion 2013-05-09 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Opiate use | 48 hours in the ICU

SECONDARY OUTCOMES:
Pain, anxiety and distress outcome measures | 48 hours in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ames, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Garnett RL, MacIntyre A, Lindsay P, Barber GG, Cole CW, Hajjar G, McPhail NV, Ruddy TD, Stark R, Boisvert D. Perioperative ischaemia in aortic surgery: combined epidural/general anaesthesia and epidural analgesia vs general anaesthesia and i.v. analgesia. Can J Anaesth. 1996 Aug;43(8):769-77. doi: 10.1007/BF03013027. PMID 8840054
- [Background] Beattie WS, Buckley DN, Forrest JB. Epidural morphine reduces the risk of postoperative myocardial ischaemia in patients with cardiac risk factors. Can J Anaesth. 1993 Jun;40(6):532-41. doi: 10.1007/BF03009738. PMID 8403120